CLINICAL TRIAL: NCT07393178
Title: High Pulse Power vs. Low Pulse Power Holmium: YAG Laser in Mini-Percutaneous Nephrolithotomy for Management of Renal Stones > 20 mm: A Randomized Controlled Trial
Brief Title: Efficacy & Safety of High Power vs. Low Power Holmium Laser in Mini-PCNL for Large Renal Stones
Acronym: miniPCNL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elghamry, Resident in urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.25.08.3291
Record Dates: First submitted 2025-12-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Renal Stones; Renal Calculi > 2 cm
Keywords: mini-PCNL; holmium-YAG; laser lithotripsy
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high power arm (Experimental): will undergo miniPCNL will high power laser setting
  Interventions: Procedure: mini percutaneous nephrolithotomy
- low power group (Placebo Comparator): will undergo miniPCNL will low power laser setting
  Interventions: Procedure: mini percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: mini percutaneous nephrolithotomy — Under fluoroscopic guidance, an 18G Chiba needle is used to access a posterior calyx or the appropriate target calyx). Contrast confirms the collecting system entry.
  Dilation is performed, typically up to 14-20 Fr. A mini-nephroscope (15 Fr) is inserted through an appropriate sheath. Irrigation is maintained using gravity or low-pressure systems.
  Holmium: YAG laser is used for lithotripsy. high pulse power will be capped at 40 W, while low pulse power settings will remain between 10-20 W. Fragments are evacuated via vacuum cleaner effect or basket through the sheath.
  Other Names: miniperc, miniPCNL

SUMMARY:
The investigator will compare between holmium laser setting during miniPCNL for renal stones as regard safety & efficacy

DETAILED DESCRIPTION:
The first 80 consecutive Patients presented to the department of urology, Mansoura Urology and Nephrology Center and fulfilling the inclusion criteria will be included in the present study.

Preoperatively, all patients will be thoroughly evaluated by medical history and physical examination including body mass index (BMI), laboratory assessment (including urine analysis/culture, serum biochemistry, CBC, bleeding profile).

Radiological assessment will include plain X-ray Kidney-Ureter-Bladder (KUB), abdominal ultrasound and non-contrast computed tomography (NCCT).

NCCT images will be obtained from above the kidneys through the bladder base. For each renal stone, location, largest diameter, burden and density will be assessed.

Culture based antibiotic is given. Under spinal anaesthesia, the patient is initially placed in lithotomy position for retrograde ureteral catheter placement, then repositioned to prone or modified supine position for percutaneous access.

Under fluoroscopic guidance, an 18G Chiba needle is used to access a posterior calyx or the appropriate target calyx). Contrast confirms the collecting system entry.

Dilation is performed, typically up to 14-20 Fr. A mini-nephroscope (15 Fr) is inserted through an appropriate sheath. Irrigation is maintained using gravity or low-pressure systems.

Holmium: YAG laser is used for lithotripsy. high pulse power will be capped at 40 W, while low pulse power settings will remain between 10-20 W. Fragments are evacuated via vacuum cleaner effect or basket through the sheath.

Depending on intraoperative findings, a nephrostomy tube and/or double-J stent may be placed. Tubeless approach may be considered.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Renal Stones < 20 mm indicated for intervention (pain, infection, obstructing stone causing hydronephrosis or parenchymal affection)
* Informed consent obtained

Exclusion Criteria:

* Active urinary tract infection
* Bleeding diathesis
* Pregnancy
* Anatomical anomalies impeding access e.g. ectopic malrotated kidneys, crossed fused kidneys...etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
operative time | during mini-PCNL procedure (intraoperative )
  time from introduction of nephroscope till nephrostomy tube fixation

SECONDARY OUTCOMES:
post operative complication | 2 days
  number of patients that will develop post operative fever, hematuria, or will require blood transfusion
stone free rate at 3 month | 3 month
  presence of residual stones requiring reintervention

IPD SHARING:
Plan to Share IPD: No